CLINICAL TRIAL: NCT04769700
Title: Post-partum Depression, Breastfeeding Adherence, and Fear in Women Giving Birth During the COVID-19 Pandemic.
Brief Title: Post-partum Depression, Breastfeeding Adherence and Fear in COVID-19
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, GONZALEZ-OJEDA ALEJANDRO, Principal Investigator, Instituto Mexicano del Seguro Social
Other Study IDs: Lactancia1
Record Dates: First submitted 2021-02-02; First posted 2021-02-24 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Breast Feeding, Exclusive; Post Partum Depression; Covid19
Keywords: COVID-19; Post-partum depression; Breast feeding; Pandemic
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum; COVID-19 | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Edinburgh Postnatal Depression Scale — The Edinburgh Postnatal Depression Scale is a self-administered questionnaire made up of 10 items scored using a four-point Likert scale (0-3) designed to screen for symptoms of postpartum depression. Postpartum depression represents the end of a continuum of severity of symptoms. The present study used a cutoff point for depressive symptomatology risk of higher than 12.
Behavioral: Breast Feeding Adherence — This will be addressed according to the breastfeeding initiation practices according to the WHO.
Behavioral: Fear of Covid-19 Scale — The Fear of Covid-19 Scale is a questionnaire that evaluates fear of the global pandemic caused by the SARS-CoV-2. It consists of seven items, each with a five-point Likert scale of options. The participant is instructed to choose the option that best represents their perception about the statement presented. The maximum possible total is 35 points. The scale's authors indicate that the higher the score is, the higher is the level of the participants' fear of COVID-19.

SUMMARY:
This study aims to explore whether quarantine measures, social distancing and hospital containment policies among women giving birth during the COVID-19 pandemic enhanced psycho-emotional distress in the immediate postpartum period. The investigators tested for depression using the Edinburgh Postnatal Depression Scale (EPDS) in the first 6 postpartum months, and then used the Fear of COVID-19 Scale, measuring also the adherence and practices of breastfeeding according to WHO.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥18 years
* Women who delivered singletons at term in the last 6 months during the COVID-19 pandemic

Exclusion Criteria:

* Women who delivered two or more products
* Women who delivered singletons at term past the last 6 months during the COVID-19 pandemic
* Women who delivered singletons pre or post-term in the last 6 months during the COVID-19 pandemic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who delivered singletons at term in the last 6 months during the COVID-19 pandemic.
Study Population: Women who delivered singletons at term in the last 6 months during the COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Post-Partum Depression Frequency | Baseline
  To explore the frequency of post-partum depression in women who gave birth during the COVID-19 pandemic
Breast Feeding Adherence and behavior. | Baseline
  To explore the breastfeeding behavior of women who gave birth during the COVID-19 pandemic. The investigators asked the patients about the frequency of breastfeeding, the duration in months of how long the mothers breastfed in a previous child, if the participants have breastfed before, and whether the participants exclusively breastfed or complemented the nutrition with formula.
Fear of Covid-19 severity | Baseline
  The Fear of Covid-19 Scale (FCV-19S) is a questionnaire that evaluates fear of the global pandemic caused by the SARS-CoV-2. The FVC-19S consists of seven items, such as "It makes me uncomfortable to think about coronavirus-19," "I am afraid of losing my life because of coronavirus-19," and "When watching news and stories about coronavirus-19 on social media, I become nervous or anxious," each with a five-point Likert scale of options. The participant is instructed to choose the option that best represents their perception about the statement presented. The maximum possible total is 35 points. The scale's authors indicate that the higher the score is, the higher is the level of the participants' fear of COVID-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano del Seguro Social, Guadalajara, Jalisco, Mexico